CLINICAL TRIAL: NCT01760941
Title: Feasibility of a Compassionate Same-Day Evaluation and Delivery of Single Fraction Radiotherapy for Palliation of Symptomatic Bony Metastasis in Hospice Patients
Brief Title: Compassionate Same-Day Evaluation & Delivery of XRT for Bony Metastasis in Hospice Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-14596; NCI-2012-03117 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Symptomatic Osseous Bone Lesions From Any Malignancy
Keywords: Urology; Prostate; Breast; Lung; Chest
MeSH Terms: interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy) (Experimental): This is a survey study to evaluate the feasibility and effectiveness of an affordable, $400 flat rate, same-day consultation, simulation, and delivery of a single fraction of palliative radiation therapy for patients with symptomatic bony metastatic disease who are currently enrolled in hospice. Treatment planning and delivery of palliative radiotherapy will utilize "standard of care" techniques. A physician survey of feasibility will be conducted on the treatment day. Patient surveys will conducted on the day of treatment and at 2 weeks, 4 weeks, 2 months, 3 months, 4 months, 5 months, and 6 months after treatment.
  Interventions: Radiation: Radiation Therapy; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: RT; Irradiation
Other: Quality-of-Life Assessment — The patient quality of life as measured by the ESAS-r; Edmonton Symptom Assessment System revised.
Other: Survey Administration — The surveys consists of Radiation Therapy Worthfullness survey; BPI: brief pain inventory; NUS: narcotics usage survey.

SUMMARY:
This is a survey study to evaluate the feasibility and effectiveness of an affordable, $400 flat rate, same-day consultation, simulation, and delivery of a single fraction of palliative radiation therapy for patients with symptomatic bony metastatic disease who are currently enrolled in hospice. Treatment planning and delivery of palliative radiotherapy will utilize "standard of care" techniques.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osseous bone lesion(s) from any malignancy, whether primary of metastatic, with histological confirmation of malignancy.
* Currently enrolled in hospice and referred for single fraction palliative radiotherapy.
* Performance status (to be evaluated by the radiation oncologist), Karnofsky Performance Scale ≥ 20 or ECOG Performance Scale < 5 .
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnancy.
* Unable to understand English.
* Unable to complete forms with assistance.
* Concurrent enrollment in a study of pain management involving medications or devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Drew Moghanaki, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiotherapy: Single fraction radiotherapy
  Radiotherapy: Single fraction radiotherapy. All study participants will be evaluated, simulated, and treated with conventional single fraction palliative radiotherapy using standard techniques with CT-based treatment.
  planning.
Period: Overall Study
Arm/Group | Radiotherapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Treatment Delivery in the Same Day as Initial Evaluation
Description: Patient evaluation will consist of surveys conducted at the time of treatment measured by the Radiation Oncologist Evaluation and Feasibility Assessments survey
Time Frame: Up to 6 months
Arm/Group | Radiotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate the Treatment Influence on the Rate of Pain Stabilization and/or Reduction
Description: Evaluate the treatment influence on the rate of pain stabilization and/or reduction as measured by the validated BPI patient questionnaire.
Time Frame: 2 weeks
Arm/Group | Radiotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Evaluate the Treatment Influence on Patient Quality of Life
Description: Evaluate the treatment influence on patient quality of life as measured by the ESAS.
Time Frame: 2 weeks
Arm/Group | Radiotherapy
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Quantify the Percentage of Patients Receiving the Treatment Who Believe That the Treatment Was Worthwhile
Description: Quantify the percentage of patients receiving the treatment who believe that the treatment was worthwhile
Time Frame: 6 months
Arm/Group | Radiotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: As this is a survey study and not a drug study, changed from an "Adverse Events" section to a "Study Risks" section. No AEs or SAEs were collected.
Arm/Group | Radiotherapy
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No data analysis or outcome measures for one participant enrolled and zero participants analyzed. Early suspension and termination due to slow accrual from Protocol Review and Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes